CLINICAL TRIAL: NCT01634113
Title: A Phase II/III, Randomised, Double-blind, Placebo-controlled, Parallel Group Trial to Evaluate Safety and Efficacy of Tiotropium Inhalation Solution (2.5 µg and 5 µg) Administered Once Daily in the Afternoon Via Respimat® Inhaler for 12 Weeks in Patients 1 to 5 Years Old With Persistent Asthma
Brief Title: Evaluation of Tiotropium 2.5 and 5 mcg Once Daily Delivered Via the Respimat® Inhaler Compared to Placebo in 1 to 5 Year Old Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.443; 2011-005512-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-04-16; First posted 2012-07-06 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (3):
- tiotropium low dose (Experimental): Once daily, delivered with Respimat® inhaler
  Interventions: Drug: tiotropium-bromide
- tiotropium high dose (Experimental): Once daily, delivered with Respimat® inhaler
  Interventions: Drug: tiotropium-bromide
- placebo (Placebo Comparator): Once daily, delivered with Respimat® inhaler
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tiotropium-bromide — IMP
  Arms: tiotropium high dose
Drug: tiotropium-bromide — IMP
  Arms: tiotropium low dose
Drug: placebo — placebo matching tiotropium
  Arms: placebo

SUMMARY:
The primary objective of this trial is to evaluate the safety and efficacy of two doses of tiotropium inhalation solution delivered via the Respimat® inhaler once daily in the afternoon in patients (1 to 5 years old) with persistent asthma on top of inhaled corticosteroid (ICS) treatment.

ELIGIBILITY:
Inclusion criteria:

1. All patients' parents (or legal guardians) must sign and date an informed consent consistent with ICH-GCP guidelines and local legislation prior to participation in the trial. Where appropriate, participants should assent to enroll in the study.
2. Male or female patients between 1 and 5 years of age.
3. By a physician documented (at least 6 month) history of persistent asthma symptoms, including (but not limited to) wheezing, cough, and/or shortness of breath. (persistent = need for inhalation corticosteroid maintenance therapy to control asthma symptoms)
4. For patients aged 5 years and capable of performing technically acceptable Pulmonary Function tests (PFTs): documented impaired lung function (i.e. pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1) is smaller or equal to 90% of predicted normal).
5. All patients must have been on maintenance treatment with an inhaled corticosteroid at stable dose, either as mono treatment or in combination with another controller medication, for at least 4 weeks before Visit 1.
6. All patients must be symptomatic (partly controlled) as defined by the Global Initiative for Asthma (GINA) guideline for children aged 5 years and younger in the week prior to Visit 1 (screening) and in the week prior to randomisation (Visit 2).

Further inclusion criteria apply.

Exclusion criteria:

1. Patients with a significant disease other than asthma.
2. Patients with clinically relevant abnormal screening haematology or blood chemistry will be excluded if the abnormality defines a significant disease as defined in exclusion criterion 1.
3. Patients with a history of congenital or acquired heart disease, or patients who have been hospitalised for cardiac syncope or failure during the past year.
4. Patients with any unstable or life-threatening cardiac arrhythmia, including cardiac arrhythmia requiring intervention (e.g. pacemaker implantation) or a change in drug therapy within the past year.
5. Patients with a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy.
6. Patients with clinically significant lung diseases other than asthma.
7. Alternative causes (other causes than asthma) that can lead to respiratory symptoms of wheeze, cough and shortness of breath.
8. Patients with known active tuberculosis.
9. Patients who have undergone thoracotomy with pulmonary resection.
10. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to the screening visit (Visit 1).

Further exclusion criteria apply.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (33):
- United States (4):
  - 205.443.12003 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 205.443.12005 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.443.12006 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.443.12004 Boehringer Ingelheim Investigational Site, Summerville, South Carolina
- Belgium (3):
  - 205.443.01004 Boehringer Ingelheim Investigational Site, Antwerp
  - 205.443.01002 Boehringer Ingelheim Investigational Site, Brussels
  - 205.443.01001 Boehringer Ingelheim Investigational Site, Edegem
- Finland (2):
  - 205.443.02002 Boehringer Ingelheim Investigational Site, Helsinki
  - 205.443.02003 Boehringer Ingelheim Investigational Site, Turku
- Germany (4):
  - 205.443.03003 Boehringer Ingelheim Investigational Site, Berlin
  - 205.443.03001 Boehringer Ingelheim Investigational Site, Bochum
  - 205.443.03002 Boehringer Ingelheim Investigational Site, Ettenheim
  - 205.443.03010 Boehringer Ingelheim Investigational Site, Frankfurt
- Latvia (3):
  - 205.443.05001 Boehringer Ingelheim Investigational Site, Balvi
  - 205.443.05003 Boehringer Ingelheim Investigational Site, Rēzekne
  - 205.443.05002 Boehringer Ingelheim Investigational Site, Riga
- Lithuania (2):
  - 205.443.06002 Boehringer Ingelheim Investigational Site, Vilnius
  - 205.443.06003 Boehringer Ingelheim Investigational Site, Vilnius
- Malaysia (3):
  - 205.443.10002 Boehringer Ingelheim Investigational Site, Kelantan
  - 205.443.10001 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.443.10003 Boehringer Ingelheim Investigational Site, Kuala Pahang
- Netherlands (2):
  - 205.443.04003 Boehringer Ingelheim Investigational Site, Breda
  - 205.443.04001 Boehringer Ingelheim Investigational Site, Groningen
- Philippines (2):
  - 205.443.09001 Boehringer Ingelheim Investigational Site, Quezon City
  - 205.443.09002 Boehringer Ingelheim Investigational Site, Quezon City
- South Korea (3):
  - 205.443.82003 Boehringer Ingelheim Investigational Site, Guri-si
  - 205.443.82002 Boehringer Ingelheim Investigational Site, Incheon
  - 205.443.82001 Boehringer Ingelheim Investigational Site, Seoul
- Ukraine (5):
  - 205.443.07003 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.443.07002 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.443.07005 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 205.443.07004 Boehringer Ingelheim Investigational Site, Zaporizhya
  - 205.443.07001 Boehringer Ingelheim Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Wachtel H, Nagel M, Engel M, El Azzi G, Sharma A, Suggett J. In vitro and clinical characterization of the valved holding chamber AeroChamber Plus(R) Flow-Vu(R) for administrating tiotropium Respimat(R) in 1-5-year-old children with persistent asthmatic symptoms. Respir Med. 2018 Apr;137:181-190. doi: 10.1016/j.rmed.2018.03.010. Epub 2018 Mar 7. PMID 29605203
- [Derived] Vrijlandt EJLE, El Azzi G, Vandewalker M, Rupp N, Harper T, Graham L, Szefler SJ, Moroni-Zentgraf P, Sharma A, Vulcu SD, Sigmund R, Chawes B, Engel M, Bisgaard H. Safety and efficacy of tiotropium in children aged 1-5 years with persistent asthmatic symptoms: a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2018 Feb;6(2):127-137. doi: 10.1016/S2213-2600(18)30012-2. Epub 2018 Jan 18. PMID 29361462

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Respimat: Inhalation of placebo solution once daily for 12 weeks, delivered by the Respimat Inhaler
- Tio R2.5: Inhalation of 2.5μg tiotropium bromide solution once daily for 12 weeks, delivered by the Respimat Inhaler
- Tio R5: Inhalation of 5μg tiotropium bromide solution once daily for 12 weeks, delivered by the Respimat Inhaler.
Period: Overall Study
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Started | 34 | 36 | 32
Completed | 34 | 36 | 31
Not Completed | 0 | 0 | 1
Not completed — Not treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set which included all randomised patients who received at least one dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5 | Total
Number analyzed (Participants) | 34 | 36 | 31 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.2 (1.4) | 3.1 (1.5) | 3.1 (1.3) | 3.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 10 | 40
  Male | 21 | 19 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Weekly Mean Combined Daytime Asthma Symptom Score
Description: Change from baseline in the weekly mean combined daytime asthma symptom score as assessed by the Paediatric Asthma Caregivers Diary (PACD) in the last week of the 12 week treatment period.
  The PACD is a diary designed to evaluate daily asthma symptoms in children aged 2-5 years. The diary consists of three questions to be answered each morning, when the child wakes up, and seven questions to be answered each evening, right after the child goes to bed for the night. A week was defined as 7 days.
  The combined daytime score is the average of scores from questions 4 - 7 in the diary which are questions regarding severity of cough, wheezing, trouble breathing and interference with activities, scores for each question range from 0 (best) to 5 (worst). The week 12 weekly mean is the mean of the responses for each day averaged over the 7 days in week 12, so combined daytime asthma symptom scores also range from 0 (best) to 5 (worst).
  The measured values presented are adjusted means.
Time Frame: Baseline and 12 weeks
Population: Full analysis set, which included all randomised patients who received at least one dose of trial medication, including patients with available endpoint data at week 12. Missing data in a week was imputed by the available data from the patient during that week, for weeks where data was completely missing no imputation was employed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 34 | 36 | 30
units on a scale | -0.456 (0.084) | -0.535 (0.082) | -0.504 (0.089)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.4963, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = -0.080, 95% CI 2-sided [-0.312 to 0.152], Standard Error of Mean 0.117 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.6936, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = -0.048, 95% CI 2-sided [-0.292 to 0.195], Standard Error of Mean 0.123 — Difference calculated as Tio R5 minus placebo

2. Primary Outcome: FEV1 Peak (0-3h) Change From Baseline
Description: Change from baseline in peak Forced expiratory volume in 1 second within the first 3 hours post dosing (FEV1 peak (0-3h)) measured at week 12
Time Frame: 10 minutes before drug administration and 30 minutes, 1 hour (h), 2h and 3h after drug administration at baseline and week 12
Population: Full analysis set including only 5 years olds capable of providing technically acceptable pulmonary function tests (PFTs). No imputation for missing data was employed.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres | 0.158 (0.026) | 0.130 (0.125) | 0.145 (0.078)

3. Secondary Outcome: Weekly Mean Overnight Asthma Symptom Score Response
Description: Change from baseline in the weekly mean overnight asthma symptom score response as assessed by the PACD in the last week of the 12 week treatment period.
  The overnight score is the score from the following question in the PACD, "How much did your child cough last night after your child was put to bed for the night until he/she awoke this morning?". This endpoint was determined only for patients with 2 or more nights with symptoms per week during the baseline period. In this case, the baseline period is the 7 days used to derive the baseline value. A patient has a night with symptoms if the question was answered with scores 1, 2, 3, 4 or 5 or the patient received β-Agonist at least one time since he/she went to bed. A week was defined as 7 days.
  Scores range from 0 (best) to 4 (worst), a value of 5 indicates severity of symptoms is unknown.
  The measured values presented are adjusted means
Time Frame: Baseline and 12 weeks
Population: Full analysis set, including patients with available endpoint data at week 12. Missing data in a week was imputed by the available data from the patient during that week, for weeks where data was completely missing no imputation was employed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 31 | 31 | 28
units on a scale | -0.671 (0.110) | -0.588 (0.111) | -0.655 (0.116)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.5995, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = 0.083, 95% CI 2-sided [-0.229 to 0.394], Standard Error of Mean 0.157 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.9251, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = 0.015, 95% CI 2-sided [-0.303 to 0.333], Standard Error of Mean 0.160 — Difference calculated as Tio R5 minus placebo

4. Secondary Outcome: Weekly Percentage of Days Without Asthma Symptoms
Description: Weekly Percentage of days without asthma symptoms at week 12.
  A day without asthma symptoms was defined as a day during which the patient experienced no asthma symptoms, did not use rescue medication (salbutamol/albuterol) and had no asthma exacerbation/worsening requiring systemic corticosteroids, or unscheduled visits to a doctor's office, emergency department, or hospital. A week was defined as 7 days.
  The measured values presented are adjusted means
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 34 | 36 | 30
percentage of days | 53.151 (7.405) | 55.401 (7.181) | 50.654 (7.873)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.8279, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = 2.250, 95% CI 2-sided [-18.243 to 22.743], Standard Error of Mean 10.324 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.8181, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = -2.497, 95% CI 2-sided [-23.987 to 18.994], Standard Error of Mean 10.826 — Difference calculated as Tio R5 minus placebo

5. Secondary Outcome: Weekly Percentage of Days With Use of Salbutamol (Albuterol) Rescue Medication
Description: Weekly percentage of days with use of salbutamol (albuterol) rescue medication at week 12. A week was defined as 7 days.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 34 | 36 | 30
percentage of days | 24.94 (36.80) | 24.23 (36.86) | 24.88 (38.45)

6. Secondary Outcome: Weekly Mean Nighttime Awakenings Due to Asthma Symptoms
Description: Change from baseline in the weekly mean nighttime awakenings due to asthma symptoms as assessed by the PACD, in the last week of the 12 week treatment period.
  The weekly mean was calculated as the average of the weekly scores for the question "Did your child wake up during the night due to his/her asthma?" The question was answered on a 5-point verbal rating scale, with scores ranging from 1 (did not wake up) to 5 (was awake all night). A week was defined as 7 days.
  The measured values presented are adjusted means
Time Frame: Baseline and 12 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 34 | 36 | 31
units on a scale | -0.318 (0.080) | -0.257 (0.078) | -0.392 (0.084)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p = 0.5869, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = 0.061, 95% CI 2-sided [-0.161 to 0.283], Standard Error of Mean 0.112 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p = 0.5230, ANCOVA — All treatment comparisons were exploratory, no formal hypothesis testing was performed; Mean Difference (Net) = -0.075, 95% CI 2-sided [-0.305 to 0.156], Standard Error of Mean 0.116 — Difference calculated as Tio R5 minus placebo

7. Secondary Outcome: Trough FEV1 Change From Baseline
Description: Change from baseline in Trough (pre-dose) Forced expiratory volume in 1 second (FEV1) measured at week 12.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres | 0.060 (0.032) | 0.017 (0.108) | 0.085 (0.163)

8. Secondary Outcome: FEV1 AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 h for FEV1 (FEV1 AUC 0-3h) after 12 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres | 0.104 (0.043) | 0.072 (0.114) | 0.077 (0.116)

9. Secondary Outcome: FVC Peak (0-3h) Change From Baseline
Description: Change from baseline in maximum forced vital capacity (FVC) measured within the first 3 hours after administration of trial medication (FVC peak (0-3h)) after 12 weeks of treatment.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres | 0.210 (0.054) | 0.136 (0.143) | 0.060 (0.085)

10. Secondary Outcome: Trough FVC Change From Baseline
Description: Change from baseline of trough (pre-dose) forced vital capacity (FVC) measured 10 min before the administration of trial medication after 12 weeks of treatment.
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres | 0.155 (0.060) | -0.027 (0.133) | -0.050 (0.226)

11. Secondary Outcome: FVC AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 h for FVC (FVC AUC0-3h) after 12 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres | 0.164 (0.037) | 0.035 (0.105) | 0.003 (0.130)

12. Secondary Outcome: Individual FEV1 Measurements
Description: Change from baseline in individual FEV1 measurements at each timepoint after 12 weeks
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres
  Time: 0 hours | 0.06 (0.03) | 0.02 (0.11) | 0.09 (0.16)
  Time: 30 minutes | 0.11 (0.09) | 0.03 (0.13) | 0.12 (0.11)
  Time: 1 hour | 0.11 (0.08) | 0.10 (0.13) | 0.12 (0.04)
  Time: 2 hours | 0.12 (0.05) | 0.09 (0.13) | 0.04 (0.16)
  Time: 3 hours | 0.10 (0.05) | 0.06 (0.13) | 0.05 (0.11)

13. Secondary Outcome: Individual FVC Measurements
Description: Change from baseline in individual FVC measurements at each timepoint after 12 weeks
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 4 | 7 | 2
Litres
  Time: 0 hours | 0.16 (0.06) | -0.03 (0.13) | -0.05 (0.23)
  Time: 30 minutes | 0.13 (0.07) | 0.04 (0.15) | 0.06 (0.08)
  Time: 1 hour | 0.18 (0.04) | 0.06 (0.14) | 0.05 (0.10)
  Time: 2 hours | 0.16 (0.04) | 0.02 (0.10) | -0.03 (0.16)
  Time: 3 hours | 0.19 (0.07) | 0.04 (0.13) | -0.03 (0.13)

ADVERSE EVENTS:
Time Frame: From first drug intake until 30 days after last drug intake, up to 119 days
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 3/34 | 0/36 | 0/31
Other Adverse Events (participants affected / at risk) | 24/34 | 19/36 | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=34) | Tio R2.5 (N=36) | Tio R5 (N=31)
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=34) | Tio R2.5 (N=36) | Tio R5 (N=31)
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1
Pyrexia (General disorders) | 6 | 3 | 3
Bronchitis (Infections and infestations) | 4 | 1 | 2
Ear infection (Infections and infestations) | 2 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 7 | 2
Pharyngitis (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 4 | 3 | 3
Rhinitis (Infections and infestations) | 3 | 2 | 3
Sinusitis (Infections and infestations) | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 5
Headache (Nervous system disorders) | 0 | 2 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.